CLINICAL TRIAL: NCT02556723
Title: Intravitreal Injections of Ziv-aflibercept for Macular Diseases: Diabetic Macular Edema, Wet AMD and Macular Edema Secondary to Vein Occlusons
Brief Title: Intravitreal Injections of Ziv-aflibercept for Macular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Retina Clinic, Sao Paulo, Brazil (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RetinaCLINIC
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Diabetic Macular Edema; Age Related Macular Degeneration; Branch Retinal Vein Occlusion With Macular Edema; Central Retinal Vein Occlusion With Macular Edema
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ziv-aflibercept IV (Experimental): All subjects will receive intravitreal injections of ziv-aflibercept under sterile conditions at baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks, and 20 weeks.
  Interventions: Drug: Intravitreal injections of ziv-aflibercept

INTERVENTIONS:
Drug: Intravitreal injections of ziv-aflibercept — All subjects will receive intravitreal injections of ziv-aflibercept under sterile conditions at baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks, and 20 weeks. No topical or systemic antibiotics will be prescribed (pre- injection or postinjection).
  Other Names: Intravitreal injections of Zaltrap

SUMMARY:
Diabetic macular edema (DME), wet-AMD and macular edema secondary to vein occlusions are the leading cause of blindness in developed countries. Several therapies have been studied as such laser treatment and intravitreal injections of corticosteroids or anti-VEGF drugs. In terms of public health the long term treatment with the current available drugs is very expensive and new therapies with the same or better effect should be investigated. This study intends to evaluate the efficacy and safety of intravitreal injections of ziv-aflibercept for the treatment of patients with DME, wet-AMD and macular edema secondary to vein occlusions.

DETAILED DESCRIPTION:
Twenty consecutive patients with DME, wet-AMD and macular edema secondary to vein occlusions will be enrolled. A complete examination including full-field ERG, visual acuity, central retinal thickness (CRT) and evaluation of systemic and ocular complications will be performed before and 24 weeks after intravitreal injections of ziv-aflibercept. The twenty patients will be submitted to 6 consecutive intravitreal injections of ziv-aflibercept with a 4 week interval.

The safety and efficacy of Eylea in the treatment of macular edema following CRVO were assessed in 2 randomized, multicenter, double- masked, sham-controlled studies: COPERNICUS and GALILEO. A total of 358 patients were treated and evaluable for efficacy (217 with Eylea) in the two studies. In both, patients were randomly assigned in a 3:2 ratio to either 2 mg Eylea administered every 4 weeks, or sham injections (control group) administered every 4 weeks for a total of 6 injections. After 6 monthly injections, patients continued to receive Eylea treatment during weeks 24 to 52 only if they met pre-specified retreatment criteria (PRN), except for patients in the sham control group in the GALILEO study who continued to receive sham injections through week 52. In the COPERNICUS study, after 6 months, 56% of patients receiving Eylea 2 mg monthly gained at least 15 letters of BCVA from baseline, as measured by ETDRS, compared to 12% of patients receiving sham injections (p<0.01), the primary endpoint of the study. Patients receiving Eylea 2 mg monthly gained, on average, 17.3 letters of vision compared to a mean loss of 4.0 letters with sham control injections (p<0.01), a secondary endpoint.

Ziv-aflibercept or zaltrap6 (Sanofi-Aventis US, LLC, Bridgewater, NJ/Regeneron Pharmaceuticals, Inc, Tarrytown, NY) is FDA approved for the treatment of metastatic colorectal cancer. During Bascom Palmer Eye Institute's Angiogenesis, Exudation, and Degeneration February 2014 conference, Michel Eid Farah, João R. Dias, Fernando M. Penha, and Eduardo B. Rodrigues investigated the safety of ziv-aflibercept in vitro and in vivo. In vitro toxicity was verified using ARPE-19 cultured cells exposed to anti-angiogenic vs balanced salt solution (BSS) for 10 minutes. Viability was assessed by 3-(4,5-dimethylthiazol-2-yl)-2,5-diphenyltetrazolium bromide (MTT) assay, which evaluates cell viability by mitochondrial activity. No signs of cell toxicity were observed, and cell viability was similar for ziv-aflibercept, aflibercept, and BSS. For the in vivo study, they tested 1 injection of 0.05 mL ziv-aflibercept vs aflibercept in the right eyes of 18 rabbits, 9 eyes in each group. BSS was injected in the fellow eyes and served as control. After the injections, all animals were examined by funduscopy, SD-OCT), and ERG at baseline, 24 hours, and 7 days. Aqueous, vitreous, and serum samples were collected at baseline, 24 hours, and 7 days for pH and osmolarity analysis. The animals were sacrificed and the eyes were enucleated for morphologic study by light and electron microscopy. No abnormalities were found at 24 hours or 7 days after intravitreal injection of either drug when assessed by fundus exam and SD-OCT, ERG, and histology as well as transmission microscopy. There were also no changes in osmolarity in the aqueous humor or vitreous samples in any group after 24 hours and 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years with type 1 or 2 diabetes mellitus
* BCVA varying from 20/62 to 20/400 (Snellen chart) - equivalent 0.49 to 1.30 logMAR - caused by DME
* Central Retinal Thickness on OCT (Heildelberg Engineering, Heidelberg, Germany ) of 275 mm or more

Exclusion Criteria:

* Laser photocoagulation within the previous 6 months
* Previous intraocular anti-VEGF or corticosteroid injection
* Previous systemic anti-VEGF or receptor tyrosine kinase inhibitor therapy
* Vitreomacular traction or epiretinal membrane producing any traction on the macula on SD-OCT scan
* Angiographic evidence of macular ischemia defined as foveal avascular zone greatest linear dimension of more than 1000 mm or severe perifoveal capillary loss
* Previous cataract, trabeculectomy or vitrectomy
* Aphakia
* External ocular infections
* Glaucoma (IOP of > 21 mmHg or regular use of more than 2 IOP lowering drugs)
* Likelihood of needing intraocular surgery within 6 months
* Proliferative diabetic retinopathy with any evidence of retinal traction
* Systemic conditions that precluded trial enrollment included glycosylated hemoglobin of more than 10.0%
* Past medical history of chronic renal failure requiring either dialysis or kidney transplantation
* Blood pressure of more than 160/90 mmHg
* an arteriothrombotic event within 6 months before randomization, including myocardial infarction, acute congestive heart failure or other cardiac event, and stroke or transient ischemic attack
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Multifocal electroretinogram responses at Week 24 and 48 | 24 and 48 weeks

SECONDARY OUTCOMES:
Change From Baseline in Best Corrected Visual Acuity (BCVA) as Measured by Snellen Letter Score at Week 24 and 48 | 24 and 48 weeks
Change From Baseline in Central Retinal Thickness (CRT) at Week 24 and 48 as Assessed on Optical Coherence Tomography (OCT) | 24 and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: André Maia, M.D., Study Director — C.E.O.
Locations (1):
- Retina Clinic / UNIFESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shaw JE, Sicree RA, Zimmet PZ. Global estimates of the prevalence of diabetes for 2010 and 2030. Diabetes Res Clin Pract. 2010 Jan;87(1):4-14. doi: 10.1016/j.diabres.2009.10.007. Epub 2009 Nov 6. PMID 19896746
- [Result] Klein R, Knudtson MD, Lee KE, Gangnon R, Klein BE. The Wisconsin Epidemiologic Study of Diabetic Retinopathy XXIII: the twenty-five-year incidence of macular edema in persons with type 1 diabetes. Ophthalmology. 2009 Mar;116(3):497-503. doi: 10.1016/j.ophtha.2008.10.016. Epub 2009 Jan 22. PMID 19167079
- [Result] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Result] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Result] Gray A, Clarke P, Farmer A, Holman R; United Kingdom Prospective Diabetes Study (UKPDS) Group. Implementing intensive control of blood glucose concentration and blood pressure in type 2 diabetes in England: cost analysis (UKPDS 63). BMJ. 2002 Oct 19;325(7369):860. doi: 10.1136/bmj.325.7369.860. PMID 12386035
- [Result] Stratton IM, Cull CA, Adler AI, Matthews DR, Neil HA, Holman RR. Additive effects of glycaemia and blood pressure exposure on risk of complications in type 2 diabetes: a prospective observational study (UKPDS 75). Diabetologia. 2006 Aug;49(8):1761-9. doi: 10.1007/s00125-006-0297-1. Epub 2006 May 31. PMID 16736131
- [Result] Ishida S, Usui T, Yamashiro K, Kaji Y, Ahmed E, Carrasquillo KG, Amano S, Hida T, Oguchi Y, Adamis AP. VEGF164 is proinflammatory in the diabetic retina. Invest Ophthalmol Vis Sci. 2003 May;44(5):2155-62. doi: 10.1167/iovs.02-0807. PMID 12714656
- [Result] Ferrara N. Vascular endothelial growth factor: basic science and clinical progress. Endocr Rev. 2004 Aug;25(4):581-611. doi: 10.1210/er.2003-0027. PMID 15294883
- [Result] Cunningham ET Jr, Adamis AP, Altaweel M, Aiello LP, Bressler NM, D'Amico DJ, Goldbaum M, Guyer DR, Katz B, Patel M, Schwartz SD; Macugen Diabetic Retinopathy Study Group. A phase II randomized double-masked trial of pegaptanib, an anti-vascular endothelial growth factor aptamer, for diabetic macular edema. Ophthalmology. 2005 Oct;112(10):1747-57. doi: 10.1016/j.ophtha.2005.06.007. PMID 16154196
- [Result] Arevalo JF, Sanchez JG, Fromow-Guerra J, Wu L, Berrocal MH, Farah ME, Cardillo J, Rodriguez FJ; Pan-American Collaborative Retina Study Group (PACORES). Comparison of two doses of primary intravitreal bevacizumab (Avastin) for diffuse diabetic macular edema: results from the Pan-American Collaborative Retina Study Group (PACORES) at 12-month follow-up. Graefes Arch Clin Exp Ophthalmol. 2009 Jun;247(6):735-43. doi: 10.1007/s00417-008-1034-x. Epub 2009 Feb 3. PMID 19189118
- [Result] Nguyen QD, Shah SM, Khwaja AA, Channa R, Hatef E, Do DV, Boyer D, Heier JS, Abraham P, Thach AB, Lit ES, Foster BS, Kruger E, Dugel P, Chang T, Das A, Ciulla TA, Pollack JS, Lim JI, Eliott D, Campochiaro PA; READ-2 Study Group. Two-year outcomes of the ranibizumab for edema of the mAcula in diabetes (READ-2) study. Ophthalmology. 2010 Nov;117(11):2146-51. doi: 10.1016/j.ophtha.2010.08.016. Epub 2010 Sep 19. PMID 20855114
- [Result] Nguyen QD, Brown DM, Marcus DM, Boyer DS, Patel S, Feiner L, Gibson A, Sy J, Rundle AC, Hopkins JJ, Rubio RG, Ehrlich JS; RISE and RIDE Research Group. Ranibizumab for diabetic macular edema: results from 2 phase III randomized trials: RISE and RIDE. Ophthalmology. 2012 Apr;119(4):789-801. doi: 10.1016/j.ophtha.2011.12.039. Epub 2012 Feb 11. PMID 22330964
- [Result] Do DV, Schmidt-Erfurth U, Gonzalez VH, Gordon CM, Tolentino M, Berliner AJ, Vitti R, Ruckert R, Sandbrink R, Stein D, Yang K, Beckmann K, Heier JS. The DA VINCI Study: phase 2 primary results of VEGF Trap-Eye in patients with diabetic macular edema. Ophthalmology. 2011 Sep;118(9):1819-26. doi: 10.1016/j.ophtha.2011.02.018. Epub 2011 May 5. PMID 21546089
- [Result] Holash J, Davis S, Papadopoulos N, Croll SD, Ho L, Russell M, Boland P, Leidich R, Hylton D, Burova E, Ioffe E, Huang T, Radziejewski C, Bailey K, Fandl JP, Daly T, Wiegand SJ, Yancopoulos GD, Rudge JS. VEGF-Trap: a VEGF blocker with potent antitumor effects. Proc Natl Acad Sci U S A. 2002 Aug 20;99(17):11393-8. doi: 10.1073/pnas.172398299. Epub 2002 Aug 12. PMID 12177445
- [Result] de Oliveira Dias JR, Badaro E, Novais EA, Colicchio D, Chiarantin GM, Matioli MM, Verna C, Penha FM, Barros NM, Meyer CH, Farah ME, Rodrigues EB. Preclinical investigations of intravitreal ziv-aflibercept. Ophthalmic Surg Lasers Imaging Retina. 2014 Nov-Dec;45(6):577-84. doi: 10.3928/23258160-20141118-15. PMID 25423640
- [Result] Mansour AM, Al-Ghadban SI, Yunis MH, El-Sabban ME. Ziv-aflibercept in macular disease. Br J Ophthalmol. 2015 Aug;99(8):1055-9. doi: 10.1136/bjophthalmol-2014-306319. Epub 2015 Feb 12. PMID 25677668
- [Result] de Oliveira Dias JR, Xavier CO, Maia A, de Moraes NS, Meyer C, Farah ME, Rodrigues EB. Intravitreal injection of ziv-aflibercept in patient with refractory age-related macular degeneration. Ophthalmic Surg Lasers Imaging Retina. 2015 Jan;46(1):91-4. doi: 10.3928/23258160-20150101-17. PMID 25559518